CLINICAL TRIAL: NCT00927901
Title: A Multi-centre, Randomized, Double-blind, Placebo-controlled, Multiple-dose, 4-way Crossover Study to Evaluate the Efficacy, Safety, Tolerability, and Pharmacokinetics of Orally Inhaled Indacaterol Salts (Maleate, Xinafoate, and Acetate) in Patients With Persistent Asthma
Brief Title: Efficacy, Safety, Tolerability, and Pharmacokinetics of Indacaterol Salts in Patients With Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CQAB149D2301; 2009-010589-46 (EudraCT Number)
Record Dates: First submitted 2009-06-24; First posted 2009-06-25 (Estimated); Results first posted 2011-08-30 (Estimated); Last update posted 2013-09-09 (Estimated); Status verified 2013-08

CONDITIONS: Asthma
Keywords: QAB149; asthma; indacaterol salts (acetate, maleate, and xinafoate); orally inhaled indacaterol salts; persistent asthma
MeSH Terms: conditions — Asthma | interventions — indacaterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- Indacaterol (ind) maleate-placebo-ind xinafoate-ind acetate (Experimental): In treatment period 1, patients received indacaterol maleate 400 μg; in treatment period 2, patients received placebo to indacaterol; in treatment period 3, patients received indacaterol xinafoate 400 μg; and in treatment period 4, patients received indacaterol acetate 400 μg. Patients received each treatment once daily for 7 days via the Concept1 single-dose dry-powder inhaler. There was a washout period of at least 7 days between each treatment period. Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short-acting β2-agonist salbutamol/albuterol was available for rescue use throughout the study.
  Interventions: Drug: Indacaterol maleate 400 μg; Drug: Indacaterol acetate 400 μg; Drug: Indacaterol xinafoate 400 μg; Drug: Placebo to indacaterol
- Indacaterol (ind) xinafoate-ind maleate-ind acetate-placebo (Experimental): In treatment period 1, patients received indacaterol xinafoate 400 μg; in treatment period 2, patients received indacaterol maleate 400 μg; in treatment period 3, patients received indacaterol acetate 400 μg; and in treatment period 4, patients received placebo to indacaterol 400 μg. Patients received each treatment once daily for 7 days via the Concept1 single-dose dry-powder inhaler. There was a washout period of at least 7 days between each treatment period. Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short-acting β2-agonist salbutamol/albuterol was available for rescue use throughout the study.
  Interventions: Drug: Indacaterol maleate 400 μg; Drug: Indacaterol acetate 400 μg; Drug: Indacaterol xinafoate 400 μg; Drug: Placebo to indacaterol
- Indacaterol (ind) acetate-ind xinafoate-placebo-ind maleate (Experimental): In treatment period 1, patients received indacaterol acetate 400 μg; in treatment period 2, patients received indacaterol xinafoate 400 μg; in treatment period 3, patients received placebo to indacaterol; and in treatment period 4, patients received indacaterol maleate 400 μg. Patients received each treatment once daily for 7 days via the Concept1 single-dose dry-powder inhaler. There was a washout period of at least 7 days between each treatment period. Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short-acting β2-agonist salbutamol/albuterol was available for rescue use throughout the study.
  Interventions: Drug: Indacaterol maleate 400 μg; Drug: Indacaterol acetate 400 μg; Drug: Indacaterol xinafoate 400 μg; Drug: Placebo to indacaterol
- Placebo-indacaterol (ind) acetate-ind maleate-ind xinafoate (Experimental): In treatment period 1, patients received placebo to indacaterol; in treatment period 2, patients received indacaterol acetate 400 μg; in treatment period 3, patients received indacaterol maleate 400 μg; and in treatment period 4, patients received indacaterol xinafoate 400 μg. Patients received each treatment once daily for 7 days via the Concept1 single-dose dry-powder inhaler. There was a washout period of at least 7 days between each treatment period. Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short-acting β2-agonist salbutamol/albuterol was available for rescue use throughout the study.
  Interventions: Drug: Indacaterol maleate 400 μg; Drug: Indacaterol acetate 400 μg; Drug: Indacaterol xinafoate 400 μg; Drug: Placebo to indacaterol

INTERVENTIONS:
Drug: Indacaterol maleate 400 μg — Indacaterol maleate 400 μg was provided in powder filled capsules with the Concept1 single-dose dry-powder inhaler. The dose refers to 400 μg of free base indacaterol.
Drug: Indacaterol acetate 400 μg — Indacaterol acetate 400 μg was provided in powder filled capsules with the Concept1 single-dose dry-powder inhaler. The dose refers to 400 μg of free base indacaterol.
Drug: Indacaterol xinafoate 400 μg — Indacaterol xinafoate 400 μg was provided in powder filled capsules with the Concept1 single-dose dry-powder inhaler. The dose refers to 400 μg of free base indacaterol.
Drug: Placebo to indacaterol — Placebo to indacaterol was provided in powder filled capsules with the Concept1 single-dose dry-powder inhaler.

SUMMARY:
This study assessed the efficacy, safety, and pharmacokinetics of indacaterol salts (maleate, xinafoate and acetate) in patients with asthma.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoker male and female adult patients aged 18-75 years inclusive, who have signed an informed consent form prior to initiation of any study-related procedure, including any adjustments to asthma medication prior to screening.
* Patients with asthma, receiving daily treatment with inhaled corticosteroid.
* Patients with a forced expiratory volume in 1 second (FEV1) during screening of ≥ 50% of the predicted normal value for the patient.
* Body mass index (BMI) must be within the range 18-32 kg/m^2 (inclusive).
* Able to communicate well with the investigator and comply with the requirements of the study.

Exclusion criteria:

* A urine cotinine level greater than the local laboratory lowest level of quantification (LOQ of 500 ng/ml or lower).
* Patients who have had a severe asthma attack/exacerbation requiring hospitalization in the 6 months prior to screening.
* Patients who have had an emergency room visit for an asthma attack/exacerbation within 6 weeks prior to screening or any time between screening and pre-dose on day 1 of the study.
* Patients who have had a respiratory tract infection within 4 weeks prior to screening or any time between screening and pre-dose on day 1 of the study.
* Patients who require the use of ≥ 8 inhalations per day of the short-acting β2-agonist salbutamol/albuterol (100 μg/90 μg salbutamol/albuterol metered dose inhaler [MDI] or equivalent dose of a dry-powder inhaler [DPI]) on any 2 consecutive days from screening to randomization.
* Patients diagnosed with chronic obstructive pulmonary disease (COPD) as defined by the Global Initiative for Chronic Obstructive Lung Disease (GOLD) guidelines (2008).
* Participation in any clinical investigation within 4 weeks prior to dosing or longer if required by local regulation. Previous participation in a study with either the investigational or comparator drugs does not exclude a patient from participation in this study.
* Significant illness.
* History of being immunocompromised, including a positive human immunodeficiency virus (HIV) test result (ELISA and Western blot).
* A positive hepatitis B surface antigen (HBsAg) or hepatitis C test result.
* Patients who are considered vulnerable as per ICH GCP guidelines.
* Patients with a history of hypersensitivity to indacaterol or to similar drugs including untoward reactions to sympathomimetic amines or inhaled medication or any component thereof.
* Treatments for asthma and allied conditions:
* The following treatments should not be used unless they have been stabilized prior to screening: antihistamines, inhaled nasal cromolyn, inhaled nasal corticosteroids, and maintenance immunotherapy.

Other protocol-defined inclusion/exclusion criteria applied to the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-06; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (3):
- Novartis Investigative Site, Poitiers, France
- Novartis Investigative Site, Wiesbaden, Germany
- Novartis Investigative Site, Verona, Italy

RESULTS

PARTICIPANT FLOW:
Groups:
- Indacaterol (Ind) Maleate-placebo-ind Xinafoate-ind Acetate: In treatment period 1, patients received indacaterol maleate 400 μg; in treatment period 2, patients received placebo to indacaterol; in treatment period 3, patients received indacaterol xinafoate 400 μg; and in treatment period 4, patients received indacaterol acetate 400 μg. Patients received each treatment for 7 days via the Concept1 single-dose dry-powder inhaler. There was a washout period of at least 7 days between each treatment period. Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short-acting β2-agonist salbutamol/albuterol was available for rescue use throughout the study.
- Indacaterol (Ind) Xinafoate-ind Maleate-ind Acetate-placebo: In treatment period 1, patients received indacaterol xinafoate 400 μg; in treatment period 2, patients received indacaterol maleate 400 μg; in treatment period 3, patients received indacaterol acetate 400 μg; and in treatment period 4, patients received placebo to indacaterol 400 μg. Patients received each treatment for 7 days via the Concept1 single-dose dry-powder inhaler. There was a washout period of at least 7 days between each treatment period. Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short-acting β2-agonist salbutamol/albuterol was available for rescue use throughout the study.
- Indacaterol (Ind) Acetate-ind Xinafoate-placebo-ind Maleate: In treatment period 1, patients received indacaterol acetate 400 μg; in treatment period 2, patients received indacaterol xinafoate 400 μg; in treatment period 3, patients received placebo to indacaterol; and in treatment period 4, patients received indacaterol maleate 400 μg. Patients received each treatment for 7 days via the Concept1 single-dose dry-powder inhaler. There was a washout period of at least 7 days between each treatment period. Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short-acting β2-agonist salbutamol/albuterol was available for rescue use throughout the study.
- Placebo-indacaterol (Ind) Acetate-ind Maleate-ind Xinafoate: In treatment period 1, patients received placebo to indacaterol; in treatment period 2, patients received indacaterol acetate 400 μg; in treatment period 3, patients received indacaterol maleate 400 μg; and in treatment period 4, patients received indacaterol xinafoate 400 μg. Patients received each treatment for 7 days via the Concept1 single-dose dry-powder inhaler. There was a washout period of at least 7 days between each treatment period. Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short-acting β2-agonist salbutamol/albuterol was available for rescue use throughout the study.
Period: Treatment Period 1
Arm/Group | Indacaterol (Ind) Maleate-placebo-ind Xinafoate-ind Acetate | Indacaterol (Ind) Xinafoate-ind Maleate-ind Acetate-placebo | Indacaterol (Ind) Acetate-ind Xinafoate-placebo-ind Maleate | Placebo-indacaterol (Ind) Acetate-ind Maleate-ind Xinafoate
Started | 7 | 7 | 7 | 9
Completed | 7 | 7 | 6 | 9
Not Completed | 0 | 0 | 1 | 0
Not completed — Subject withdrew consent | 0 | 0 | 1 | 0
Period: Treatment Period 2
Arm/Group | Indacaterol (Ind) Maleate-placebo-ind Xinafoate-ind Acetate | Indacaterol (Ind) Xinafoate-ind Maleate-ind Acetate-placebo | Indacaterol (Ind) Acetate-ind Xinafoate-placebo-ind Maleate | Placebo-indacaterol (Ind) Acetate-ind Maleate-ind Xinafoate
Started | 7 | 7 | 6 | 9
Completed | 7 | 7 | 6 | 9
Not Completed | 0 | 0 | 0 | 0
Period: Treatment Period 3
Arm/Group | Indacaterol (Ind) Maleate-placebo-ind Xinafoate-ind Acetate | Indacaterol (Ind) Xinafoate-ind Maleate-ind Acetate-placebo | Indacaterol (Ind) Acetate-ind Xinafoate-placebo-ind Maleate | Placebo-indacaterol (Ind) Acetate-ind Maleate-ind Xinafoate
Started | 7 | 7 | 6 | 9
Completed | 7 | 7 | 6 | 9
Not Completed | 0 | 0 | 0 | 0
Period: Treatment Period 4
Arm/Group | Indacaterol (Ind) Maleate-placebo-ind Xinafoate-ind Acetate | Indacaterol (Ind) Xinafoate-ind Maleate-ind Acetate-placebo | Indacaterol (Ind) Acetate-ind Xinafoate-placebo-ind Maleate | Placebo-indacaterol (Ind) Acetate-ind Maleate-ind Xinafoate
Started | 7 | 7 | 6 | 9
Completed | 7 | 7 | 5 | 8
Not Completed | 0 | 0 | 1 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1
Not completed — Subject withdrew consent | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: The entire study population included all 4 treatment groups who received the 3 salt forms of indacaterol 400 µg (maleate, acetate, and xinafoate) and placebo to indacaterol in 4 different sequences. The dose refers to 400 μg of free base indacaterol. Patients received each treatment for 7 days via the Concept1 single-dose dry-powder inhaler. There was a washout period of at least 7 days between each treatment period. Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short-acting β2-agonist salbutamol/albuterol was available for rescue use throughout the study.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 30
Age Continuous [Mean (Standard Deviation); unit: years] | 50 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 23

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Trough Forced Expiratory Volume in 1 Second (FEV1) 24 Hours Post-dose at the End of Each Treatment Period (Day 7)
Description: FEV1 was measured with spirometry conducted according to internationally accepted standards. Trough FEV1 was defined as the average of measurements made 23 hours 10 minutes and 23 hours 45 minutes post-dose at Baseline and at the end of each treatment period. The analysis included period baseline FEV1 as covariate.
Time Frame: Baseline to the end of each treatment period (Day 7)
Population: Efficacy analysis set: All randomized subjects that received at least 1 dose of study drug and had a baseline and at least 1 post-baseline measurement of FEV1.
Measure: Least Squares Mean (90% Confidence Interval); unit: Liters
Groups:
- Indacaterol Maleate 400 μg: Patients received indacaterol maleate 400 μg once daily for 7 days via the Concept1 single-dose dry-powder inhaler. The dose refers to 400 μg of free base indacaterol. Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short-acting β2-agonist salbutamol/albuterol was available for rescue use throughout the study.
- Indacaterol Acetate 400 μg: Patients received indacaterol acetate 400 μg once daily for 7 days via the Concept1 single-dose dry-powder inhaler. The dose refers to 400 μg of free base indacaterol. Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short-acting β2-agonist salbutamol/albuterol was available for rescue use throughout the study.
- Indacaterol Xinafoate 400 μg: Patients received indacaterol xinafoate 400 μg once daily for 7 days via the Concept1 single-dose dry-powder inhaler. The dose refers to 400 μg of free base indacaterol. Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short-acting β2-agonist salbutamol/albuterol was available for rescue use throughout the study.
- Placebo to Indacaterol: Patients received placebo to indacaterol once daily for 7 days via the Concept1 single-dose dry-powder inhaler. Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short-acting β2-agonist salbutamol/albuterol was available for rescue use throughout the study.
Arm/Group | Indacaterol Maleate 400 μg | Indacaterol Acetate 400 μg | Indacaterol Xinafoate 400 μg | Placebo to Indacaterol
Number analyzed (Participants) | 28 | 29 | 28 | 29
Liters | 0.186 [0.1079 to 0.2649] | 0.190 [0.1133 to 0.2673] | 0.194 [0.1164 to 0.2728] | -0.021 [-0.0982 to 0.0558]

2. Secondary Outcome: Change From Baseline in Trough Forced Expiratory Volume in 1 Second (FEV1) 24 Hours Post-dose on Day 1
Description: FEV1 was measured with spirometry conducted according to internationally accepted standards. Trough FEV1 was defined as the average of measurements made 23 hours 10 minutes and 23 hours 45 minutes post-dose at Baseline and on Day 1. The analysis included period baseline FEV1 as covariate.
Time Frame: Baseline to Day 1
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: Liters
Arm/Group | Indacaterol Maleate 400 μg | Indacaterol Acetate 400 μg | Indacaterol Xinafoate 400 μg | Placebo to Indacaterol
Number analyzed (Participants) | 29 | 30 | 29 | 29
Liters | 0.161 [0.0877 to 0.2344] | 0.185 [0.1129 to 0.2572] | 0.205 [0.1325 to 0.2792] | 0.008 [-0.0649 to 0.0819]

3. Secondary Outcome: Time to Peak Forced Expiratory Volume in 1 Second (FEV1) on Day 1 and Day 7
Description: FEV1 was measured with spirometry conducted according to internationally accepted standards at 5, 15, and 30 minutes; 1 hour, 1 hour 30 minutes; and 2, 4, and 12 hours post-dose on Day 1 and Day 7.
Time Frame: Day 1 and Day 7
Population: as for outcome 1
Measure: Median (90% Confidence Interval); unit: Hours
Arm/Group | Indacaterol Maleate 400 μg | Indacaterol Acetate 400 μg | Indacaterol Xinafoate 400 μg | Placebo to Indacaterol
Number analyzed (Participants) | 29 | 30 | 29 | 29
Hours
  Day 1, N=29, 30, 29, 29 | 4.00 [3.000 to 6.125] | 2.13 [1.500 to 3.000] | 1.50 [1.040 to 2.500] | 2.25 [1.500 to 12.085]
  Day 7, N=28, 29, 28, 29 | 3.00 [2.000 to 4.000] | 2.50 [1.500 to 4.000] | 3.00 [1.250 to 12.000] | 12.38 [11.710 to 13.875]

4. Secondary Outcome: Percentage of Patients Using Rescue Medication During Each 7 Day Treatment Period
Description: Patients recorded use of rescue medication (salbutamol/albuterol multi-dose inhaler) as the number of puffs taken in respective preceding 12 hours morning and evening in a diary. Patient with any use of rescue medication (any number of puffs > 0) was included to calculate endpoint.
Time Frame: Baseline to the end of each treatment period (Day 7)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Groups:
- Indacaterol Acetate 400 μg: 3Patients received indacaterol acetate 400 μg once daily for 7 days via the Concept1 single-dose dry-powder inhaler. The dose refers to 400 μg of free base indacaterol. Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short-acting β2-agonist salbutamol/albuterol was available for rescue use throughout the study.
Arm/Group | Indacaterol Maleate 400 μg | Indacaterol Acetate 400 μg | Indacaterol Xinafoate 400 μg | Placebo to Indacaterol
Number analyzed (Participants) | 29 | 30 | 29 | 29
Percentage of participants | 21 | 10 | 17 | 21

5. Secondary Outcome: Indacaterol Exposure (AUC[0-24 Hours]) at the End of Each 7 Day Treatment Period
Description: Venous blood samples for pharmacokinetic evaluation were collected at 15 and 30 minutes; and 1, 2, 4, 12, and 24 hours post-dose at the end of each 7 day treatment period and were analyzed using a LC-MS/MS assay. Area under the concentration-time curve up to 24 hours (AUC[0-24 hours]) was calculated from concentration-time data and recorded sampling times using non-compartmental methods.
Time Frame: End of each treatment period (Day 7)
Population: Pharmacokinetic analysis set: All subjects with evaluable pharmacokinetic parameter data. Number of subjects varied due to missing values.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg * hr/mL
Arm/Group | Indacaterol Acetate 400 μg | Indacaterol Maleate 400 μg | Indacaterol Xinafoate 400 μg
Number analyzed (Participants) | 29 | 28 | 27
pg * hr/mL | 5159 (27.9) [3003 to 10893] | 5434 (30.7) [3581 to 13634] | 5170 (24.2) [3312 to 8349]

6. Secondary Outcome: Indacaterol Exposure (Cmax) at the End of Each 7 Day Treatment Period
Description: Venous blood samples for pharmacokinetic evaluation were collected at 15 and 30 minutes; and 1, 2, 4, 12, and 24 hours post-dose at the end of each 7 day treatment period and were analyzed using a LC-MS/MS assay. Maximum (peak) plasma drug concentration after drug administration (Cmax) was calculated from concentration-time data and recorded sampling times using non-compartmental methods.
Time Frame: End of each treatment period (Day 7)
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | Indacaterol Acetate 400 μg | Indacaterol Maleate 400 μg | Indacaterol Xinafoate 400 μg
Number analyzed (Participants) | 28 | 28 | 28
pg/mL | 720 (35.5) [338 to 1550] | 753 (40.6) [322 to 1870] | 664 (26.4) [397 to 1150]

ADVERSE EVENTS:
Time Frame: Baseline to the end of the study (approximately 11 weeks)
Description: Safety population: All subjects who received at least 1 dose of study drug.
Arm/Group | Indacaterol Acetate 400 μg | Indacaterol Maleate 400 μg | Indacaterol Xinafoate 400 μg | Placebo to Indacaterol
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/29 | 0/29 | 0/29
Other Adverse Events (participants affected / at risk) | 5/30 | 4/29 | 7/29 | 5/29
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Indacaterol Acetate 400 μg (N=30) | Indacaterol Maleate 400 μg (N=29) | Indacaterol Xinafoate 400 μg (N=29) | Placebo to Indacaterol (N=29)
Nasopharyngitis (Infections and infestations) | 0 | 0 | 4 | 1
Headache (Nervous system disorders) | 1 | 1 | 2 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.